CLINICAL TRIAL: NCT01056471
Title: Multicenter Clinical Trial Phase I / II Randomized, Placebo-controlled Study to Evaluate Safety and Feasibility of Therapy With Two Different Doses of Autologous Mesenchymal Stem Cells in Patients With Secondary Progressive Multiple Sclerosis Who do Not Respond to Treatment
Brief Title: Autologous Mesenchymal Stem Cells From Adipose Tissue in Patients With Secondary Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMM/EM/2008
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-02

CONDITIONS: Autoimmune Diseases; Immune System Diseases; Demyelinating Diseases; Nervous System Diseases; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System
Keywords: Multiple Sclerosis; Mesenchymal Stem Cells; Autologous
MeSH Terms: conditions — Autoimmune Diseases; Immune System Diseases; Demyelinating Diseases; Nervous System Diseases; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose autologous mesenchymal cells (Experimental): The dose of infused cells is 10e6 cells/Kg
  Interventions: Other: Autologous mesenchymal stem cells from adipose tissue.
- High dose (Experimental): The dose of infused cells is 4*10e6 cells/Kg
  Interventions: Other: Autologous mesenchymal stem cells from adipose tissue.
- Placebo Control (No Intervention)

INTERVENTIONS:
Other: Autologous mesenchymal stem cells from adipose tissue. — Intravenous infusion of autologous mesenchymal stem cells.Dose:4*10e6 cells/Kg.
  Arms: High dose
Other: Autologous mesenchymal stem cells from adipose tissue. — Intravenous infusion of autologous mesenchymal stem cells. Dose: 10e6 cells/Kg.
  Arms: Low dose autologous mesenchymal cells

SUMMARY:
The main purpose of this study is to evaluate the safety and feasibility of regenerative therapy with mesenchymal stem cells from adipose tissue, administered intravenously in patients with secondary progressive multiple sclerosis who do not respond to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Multiple Sclerosis (Poser and McDonald criteria).
2. Secondary progressive MS patients with EDSS ≥ 5.5 and ≤ 9.
3. Patients with treatment failure defined by: no response to immunomodulators / immunosuppressants, and showing activity in the form of 1 relapse in the last year or 0.5 points in EDSS progression.
4. Patients with no MS relapse and no steroid treatment within the month prior to inclusion.
5. Patients who give written consent to participate in the study. -

Exclusion Criteria:

1. History of current pathology or current laboratory results indicative of any severe disease.
2. Pacemaker or metallic implants that prevent MR imaging.
3. Inability to complete questionnaires.
4. Refusal to give informed consent.
5. Predicted impossibility for a biopsy of at least 30 grams of fat tissue.
6. Positive screening test for HIV, Hepatitis B or Hepatitis C.
7. History of malignancy.
8. Having been in treatment with any investigational drug or have undergone any experimental procedure in the 3 months prior to baseline.
9. Body mass index> 40 kg/m2.
10. Patients who have been treated with prohibited concomitant medication during the month prior to inclusion in the study.
11. Pregnancy or lactation

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability related to the intravenous infusion of autologous mesenchymal stem cells | 12 months.

SECONDARY OUTCOMES:
To evaluate effects on MS disease activity measured by: clinical variables, imaging variables, immunological and neurophysiologic analysis, neuropsychological and quality of life scales. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Fernandez Fernandez, MD, PhD, Study Director — Hospital Regional Universitario Carlos Haya, Málaga, Spain.; Guillermo Izquierdo Ayuso, MD, PhD, Principal Investigator — Hospital Universitario Virgen Macarena, Sevilla, Spain
Locations (2):
- Spain (2):
  - Hospital Regional Universitario de Málaga, Málaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville, Sevilla

REFERENCES:
- See also: Andalusian Molecular Biology and Regenerative Medicine Centre — http://www.cabimer.es